CLINICAL TRIAL: NCT00399464
Title: Efficacy and Safety of SL77.0499-10 10mg Once Daily in Comparison With Placebo and Tamsulosin Hydrochloride 0.2mg in Patients With Lower Urinary Tract Symptoms Related to Benign Prostatic Hyperplasia (BPH).
Brief Title: Efficacy and Safety of SL77.0499-10 (Alfuzosin) Versus Placebo and Tamsulosin in Japanese Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5791
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Adrenergic alpha-Antagonists; alfuzosin
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: alfuzosin

SUMMARY:
The primary objective of the study is to demonstrate the superiority of SL77.0499-10 10mg once daily over placebo and the non-inferiority versus tamsulosin hydrochloride after 12 weeks treatment in terms of the efficacy in patients with lower urinary tract symptoms related to BPH.

The secondary objective is to assess the safety of SL77.0499-10 in patients with lower urinary tract symptoms related to BPH in comparison with placebo and tamsulosin hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Japanese;
* Having a symptomatic BPH diagnosed clinically by digital rectal examination and ultrasonography within the last 6 months;
* Suffering for at least 6 months from lower urinary tract symptoms related to BPH.

Exclusion Criteria:

* Patients with mental disorders or who cannot be relied upon to understand the trial requirements and comply with the treatment regiment;
* Inpatient;
* Patients having participated in a clinical trial within the previous 6-month;
* Patients previously treated with SL77.0499-10;
* Patients whose I-PSS total score do not meet ≥ 13;
* Patients whose urinary peak flow rate (PFR) do not meet 5.0-12.0mL/s for a voided volume of at least 150mL;
* Patients whose residual urine are > 200mL;

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in I-PSS (International Prostate Symptom Score) total score from baseline to endpoint (Day 84 or last available post-baseline assessment)

SECONDARY OUTCOMES:
Efficacy: Change in I-PSS total score from baseline to each visit
Change in Quality Of Life score from baseline to each visit
Change from baseline to endpoint of residual urine volume and urinary Peak Flow
Safety:Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan